CLINICAL TRIAL: NCT07007104
Title: Exploring the Impact of Mindful Eating: A Pilot Study Among Breast Cancer Survivors in Türkiye
Brief Title: Mindful Eating in Breast Cancer Survivors: A Pilot Study in Türkiye
Acronym: MIND-BR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Collaborators: Acibadem Altunizade Hospital, Istanbul (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-CancerStudy
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Survivorship; Eating Behavior; Weight Management; Mindful Eating Intervention
Keywords: Behavioral intervention; Breast cancer survivors; Eating behavior; Intuitive eating; Mindful eating; Weight management
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Eating Intervention + Treatment as Usual (MEI + TAU) (Experimental): Participants in this group received six structured sessions of a mindful eating intervention over a defined period, each lasting 60-90 minutes. The intervention was delivered by a registered dietitian certified in both Mindful Eating Certificate (The Center of Mindful Eating, EatRight Certified, 2023) and Mindfulness-Based Eating Awareness Training (MB-EAT) (Mindful Eating Training Institute, 2019). These sessions aimed to improve awareness of hunger and satiety cues, reduce emotional eating, and promote healthier eating behaviors. In addition to the behavioral sessions, participants also received standard post-treatment care, including individualized nutritional counseling by an oncology dietitian.
  Interventions: Behavioral: Mindful Eating Intervention; Behavioral: Oncology Nutrition Counseling
- Treatment as Usual (TAU) (Active Comparator): Participants in this group received standard survivorship care, which included individualized nutritional education and counseling delivered by an oncology dietitian. They did not participate in any mindful eating-specific behavioral intervention. This group served as the comparator to evaluate the added effect of the structured mindful eating program.
  Interventions: Behavioral: Oncology Nutrition Counseling

INTERVENTIONS:
Behavioral: Mindful Eating Intervention — The mindful eating intervention consisted of six structured group sessions delivered over a six-week period, each lasting approximately 60-90 minutes. The sessions were led by a registered dietitian certified in both Mindful Eating (The Center of Mindful Eating, EatRight Certified, 2023) and Mindfulness-Based Eating Awareness Training (MB-EAT, 2019). The curriculum was designed to improve participants' awareness of hunger and satiety cues, reduce emotional eating, enhance eating satisfaction, and foster non-judgmental eating practices. Each session incorporated guided mindfulness practices, cognitive-behavioral techniques, and experiential activities such as sensory-focused eating. The intervention was provided in addition to standard post-treatment care, which included nutritional counseling by an oncology dietitian.
  Arms: Mindful Eating Intervention + Treatment as Usual (MEI + TAU)
Behavioral: Oncology Nutrition Counseling — Participants in this group received individualized nutrition counseling and education from a registered oncology dietitian as part of standard post-treatment care for breast cancer survivors. The counseling focused on balanced eating, long-term weight management, and general lifestyle guidance based on survivorship needs. No additional behavioral or mindful eating interventions were delivered.

SUMMARY:
The goal of this clinical trial is to explore whether a mindful eating intervention can improve eating behaviors and support sustainable weight management among female breast cancer survivors in Türkiye who have completed active treatment.

The main questions it aims to answer are:

* Can a structured mindful eating program improve intuitive and mindful eating behaviors?
* Does the intervention lead to favorable changes in body weight, BMI, waist circumference, and fat mass compared to usual care?

Researchers will compare a group receiving a 6-session mindful eating intervention plus treatment-as-usual (MEI + TAU) to a treatment-as-usual (TAU) control group to see if the intervention provides additional benefits on eating behaviors and body composition.

Participants will:

* Attend six 60-90 minute group sessions on mindful eating delivered by trained professionals
* Receive tailored nutrition education from an oncology dietitian
* Complete validated questionnaires (IES-2 and MEQ-30) and anthropometric assessments at baseline and follow-up

DETAILED DESCRIPTION:
This randomized controlled pilot study investigates the effects of a six-session mindful eating intervention (MEI) on eating behaviors and body composition among female breast cancer (BC) survivors in Türkiye. Participants were recruited from a medical oncology clinic and were eligible if they had completed surgery, chemotherapy, and radiotherapy, with or without ongoing hormone therapy, at least six months prior to enrollment. A total of 25 participants were randomly assigned to one of two groups: (1) MEI combined with treatment-as-usual (MEI + TAU, n = 12) and (2) treatment-as-usual alone (TAU, n = 13).

The MEI consisted of six weekly 60-90 minute sessions led by a trained mindful eating facilitator and a registered dietitian with oncology experience. Sessions addressed themes such as recognizing hunger and satiety cues, slowing down during meals, managing emotional eating, and enhancing sensory awareness. Participants also received individualized nutritional counseling based on their anthropometric data and dietary habits.

Data were collected at baseline and multiple follow-up points across six months. Outcomes included body weight, BMI, waist circumference, fat mass, and scores from two validated behavioral questionnaires: the Intuitive Eating Scale-2 (IES-2) and the Mindful Eating Questionnaire-30 (MEQ-30). Body composition was assessed using bioelectrical impedance analysis (BIA), and statistical analysis was performed to evaluate within-group and between-group changes over time.

Preliminary results suggest that participants in the MEI + TAU group experienced significant improvements in intuitive eating scores, particularly in reliance on hunger/satiety cues and reduced emotional eating. Mindful eating scores also increased across several subscales, and reductions in waist circumference were more pronounced in the intervention group. These findings indicate that mindful eating interventions may support sustainable weight management and improved eating behaviors in breast cancer survivors. Further large-scale studies are warranted to confirm these outcomes and explore long-term effects on survivorship and recurrence risk.

ELIGIBILITY:
Inclusion Criteria:

* Female individuals aged 18 years and older
* History of breast cancer diagnosis (any subtype)
* Completion of active cancer treatment (surgery, chemotherapy, and/or radiotherapy) at least 6 months prior to enrollment
* Ability to participate in group-based behavioral sessions
* Ability to provide informed consent

Exclusion Criteria:

* Completion of cancer treatment less than 6 months prior to enrollment
* Presence of metastatic disease or active cancer recurrence
* Concurrent diagnosis of another major illness affecting dietary behavior (e.g., eating disorder, severe gastrointestinal disease)
* Cognitive impairment or psychiatric condition that limits ability to participate in behavioral sessions
* Inability or unwillingness to attend group intervention sessions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Change in Intuitive Eating Score (IES-2 Total) | Baseline and 6 months post-intervention
  The Intuitive Eating Scale-2 (IES-2) is a validated tool measuring reliance on internal cues and rejection of dieting. Higher scores reflect greater intuitive eating behavior.
Change in Mindful Eating Score (MEQ-30 Total) | Baseline and 6 months post-intervention
  The MEQ-30 evaluates domains such as awareness, emotional eating, disinhibition, and responsiveness to hunger cues. Higher scores indicate stronger mindful eating behaviors.

SECONDARY OUTCOMES:
Change in Body Fat Mass (kg) | Baseline and 6 months
  Fat mass was assessed using bioelectrical impedance analysis (BIA, Tanita MC780). Measurements were taken during individual sessions with an oncology dietitian at baseline and after 6 months.
Change in Fat-Free Mass (kg) | Baseline and 6 months
  Fat-free mass (lean mass) was measured by BIA during dietitian-led consultations.
Change in Waist Circumference (cm) | Baseline and 6 months
  Waist circumference was measured using standardized tape during sessions with an oncology dietitian to assess changes in central adiposity.

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem Altunizade Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and ethical restrictions. The current study was approved under conditions that limit data use to the research team, and participant-level data were not collected with explicit consent for external sharing. Group-level findings will be reported in scientific publications.